CLINICAL TRIAL: NCT06690151
Title: CATAMARAN - Neonatal Cohort : Characterization and Support of Neurodevelopmental Disorders Associated With Congenital Cardiac malfoRmations - Neonatal
Brief Title: Characterization and Support of Neurodevelopmental Disorders Associated With Congenital Cardiac malfoRmations - Neonatal
Acronym: CATAMARAN - NN
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Pays de la Loire Laboratory of Psychology (LPPL) (Unknown); Physiopathology of Nutritional Adaptations Joint Research Unit (UMR PhAN) (Unknown); Institut du thorax, INSERM UMR1087 (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC23_0547; IDRCB (ANSm) : 2024-A00425-42 (Other: Agence nationale de sécurité du médicament et des produits de santé (ANSM))
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Heart Disease Congenital; Neurodevelopmental Disorder
Keywords: Congenital heart defects (CHD); neurodevelopmental disorders (NDD); genetics
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders | interventions — Data Collection; Blood Circulation; Prenatal Care; Pregnancy; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Infant blood sample
  * Infant stool collection
  * Paternal blood sample
  * Maternal blood sample
  * Umbilical cord venous blood sample
  * Meconium
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study population (Newborns with congenital heart defects and their two parents): The study population will consist of 150 fetuses with a prenatally diagnosed critical congenital heart defect (CHD), at high risk of developing developmental delays, and their two parents.
  Interventions: Behavioral: Neurodevelopmental assessment (Bayley-IV); Other: Biological sampling; Behavioral: ELFE dietary questionnaire; Behavioral: Post-Traumatic Stress Questionnaire IES-R (Impact of Event Scale - Revised); Other: Data collection for the study (Cardiovascular, developemental, fetal, pregnancy, MRI)

INTERVENTIONS:
Behavioral: Neurodevelopmental assessment (Bayley-IV) — Assessment of developmental delays through administration of the Bayley-4 test by a neuropsychologist
Other: Biological sampling — The samples to be collected at delivery will include:
  * A 4 ml maternal blood sample in an EDTA tube for lipidomic and metabolomic analyses at delivery
  * A 6 ml maternal blood sample in an EDTA tube (2 tubes of 3 ml) for genetic analysis
  * A 4 ml venous cord blood sample in an EDTA tube for transcriptomic and epigenetic analysis; and a 2 ml EDTA tube for metabolomic/lipidomic analysis
  * Samples from fresh placenta for transcriptomic, epigenetic, metabolomic, and lipidomic analyses
  * A meconium sample collected as soon as possible after birth in a dry tube for microbiome analysis
  During hospitalization for the cardiac surgery:
  * Genome analysis samples will be collected from the father and the infant. These samples will be taken in two EDTA tubes of 3 ml each.
  * Perioperative neurobiomarker samples will be collected (one EDTA tube of 500 μL preoperatively and postoperatively on Day 1 and 2).
  At 1 month, a stool sample will be collected from the infants for microbiome analysis.
Behavioral: ELFE dietary questionnaire — Questionnaire on diet and lifestyle during pregnancy (only for the mother)
Behavioral: Post-Traumatic Stress Questionnaire IES-R (Impact of Event Scale - Revised) — The IES-R is a 22-item self-report measure (for DSM-IV) that assesses subjective distress caused by traumatic events.
Other: Data collection for the study (Cardiovascular, developemental, fetal, pregnancy, MRI) — * Cardiovascular follow-up data collection
  * Developmental follow-up data collection
  * Collection of postoperative brain MRI data, scheduled between Day 5 post-surgery and the end of the hospital stay
  * Collection of data on pregnancy exposure, obstetric events, and delivery data.
  * Collection of fetal ultrasound data (T2 and T3).
  * Collection of fetal echocardiography data (T2 and T3).

SUMMARY:
Congenital heart defects (CHD), as the leading cause of birth defects, affect 12 million people globally and approximately 41,000 newborns each year in Europe. CHD presents a significant public health concern due to its association with high morbidity and mortality rates across the lifespan. Over 50% of infants born with critical CHD will develop neurodevelopmental disorders (NDD), requiring specialized care and impacting their quality of life. NDDs, involving early and persistent disruptions in cognitive, emotional, and behavioral development due to abnormal brain development, are highly variable. They may impact language, learning, motor skills, intellectual efficiency, social cognition, attention, memory, and executive functions, often accompanied by psychosocial difficulties. These hidden disabilities constitute the primary long-term sequelae of CHD, surpassing even cardiovascular complications in impact, and affect children who often undergo multiple cardiac surgeries during early childhood. NDDs are associated not only with complex CHDs but also with simpler CHDs that are repaired in early childhood and considered 'cured.'

The origin of CHD-associated NDDs remains largely unknown. While few genetic or environmental causes have been identified, recent research suggests a possible common origin linking heart malformations and neurodevelopmental abnormalities. The CATAMARAN neonatal cohort project aims to detect developmental delays associated with CHD as early as six months of age and to identify both individual susceptibility factors and acquired vulnerabilities contributing to the development of NDDs in infants with CHD.

ELIGIBILITY:
The inclusion criteria are as follows:

* Fetus with a congenital heart defect (CHD) detected prenatally (prenatal diagnosis of the heart defect)
* Fetus with a critical CHD defined as requiring cardiac surgery during the first three months of the infant's life
* Parents affiliated with or beneficiaries of a social security or equivalent system
* Parents' good understanding of the French language
* Voluntary, informed, and written consent from both parents for themselves and the unborn child

Criteria for parents*:

- Biological parents *The inclusion of the father in the project does not limit the participation of the child (patient) in the study.

*The father will be encouraged to participate in the project by providing a blood sample to create a trio (mother/father/infant) for future genetic analyses.

However, if the father is unavailable or does not consent to the collection and storage of samples for analysis (as part of the CATAMARAN study or future research projects related to biobanking), the child can still be included in the study.

Exclusion Criteria:

* Medical termination of pregnancy considered
* Genetic anomaly or malformative syndrome identified prior to inclusion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will focus on the inclusion of 150 fetuses with a prenatally diagnosed critical congenital heart defect (CHD), at high risk of developing developmental delays, and their two parents.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2027-08-28 (Estimated); Study Completion 2027-08-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the prevalence of developmental delays in infants with a critical congenital heart defect (CHD) at 6 months of age. | 6 months

SECONDARY OUTCOMES:
Evaluate the prevalence of developmental delay in infants with congenital heart defects (CHD) based on the type of heart defect. | 6 months
Assess the presence of developmental delay in infants with CHD based on the complexity of cardiac surgery. | 6 months
Evaluate and describe affected developmental domains. | 6 months
Identify rare genetic variants associated with developmental delays in CHD patients through genome-wide analysis. | 6 months
Identify common genetic variants associated with developmental delays in CHD patients through genome-wide analysis. | 6 months
Characterize placental anatomopathological anomalies in CHD and their correlation with developmental delay at 6 months. | 6 months
Determine maternal dietary habits during the third trimester, their correlation with placental anomalies, and developmental delay at 6 months. | 6 months
Characterize maternal behavioral exposures (e.g., tobacco, alcohol, drugs) and obstetric complications (e.g., hypertension, preeclampsia, gestational diabetes) during pregnancy, and their correlation with placental anomalies and developmental delay | 6 months
Characterize antenatal determinants of developmental delay through multi-omics analysis (metabolomics, lipidomics, transcriptomics, and epigenetics) of maternal blood, placental function, and fetal blood, and their correlation with developmental delay | 6 months
Characterize neonatal microbiota and its association with developmental delay at 6 months. | 6 months
Identify perioperative determinants of developmental delay in CHD. | 6 months
Identify optimal perfusion pressure targets during and after neonatal cardiac surgery under cardiopulmonary bypass in three participating centers using continuous analysis of invasive blood pressure and cerebral oxygen saturation | up to 3 months
For CHU Nantes patients only: identify fetal neuronal biomarkers at birth, track their evolution before and after cardiac surgery in CHD infants, and establish associations with developmental delay at 6 months. | 6 months
Evaluate parental post-traumatic stress at 1) antenatal inclusion, 2) perioperative period, and 3) 6 months post-surgery, and its correlation with developmental delay at 6 months. | 6 months

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Nantes University Hospital, Nantes, Loire Atlantique
  - AP-HM, Marseille
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided